CLINICAL TRIAL: NCT02054390
Title: Angiotensin Converting Enzyme Inhibitor Therapy and Periprocedural Myocardial Infarction in Patients With Metabolic Syndrome
Brief Title: Angiotensin Converting Enzyme Inhibitors and Periprocedural Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Özgür Ulaş Özcan, MD, Ankara University
Other Study IDs: ACEmetsend
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Metabolic Syndrome; Coronary Artery Disease
Keywords: Angiotensin converting enzyme inhibitor; inflammation; metabolic syndrome; myonecrosis; percutaneous coronary intervention; periprocedural myocardial injury
MeSH Terms: conditions — Metabolic Syndrome; Coronary Artery Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Metabolic syndrome (MS) has been reported as a risk for cardiovascular events. The aim of the present cohort study is to investigate whether ACEi therapy reduces the rate of periprocedural myocardial injury (PPMI) after elective percutaneous coronary intervention (PCI) among patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. metabolic syndrome
2. elective percutaneous coronary intervention with angiographically successful stent implantation

Exclusion Criteria:

1. acute coronary events
2. renal failure
3. needed the use of IV glycoprotein IIb/IIIa receptor inhibitors were excluded
4. left main coronary artery disease
5. chronic total occlusion
6. high levels of baseline CKMB or troponin
7. any contraindication of aspirin, clopidogrel or ACEi treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metabolic syndorme (MS) was defined as the presence of 3 or more of these components:
  1. high fasting glucose (fasting serum glucose ≥100 mg/dl or drug treatment for elevated blood glucose)
  2. abdominal obesity (given as waist circumference >102 cm in men and >88 cm in women)
  3. high blood pressure (>130/>85 mmHg or drug treatment for hypertension)
  4. hypertriglyceridemia (serum triglycerides ≥150 mg/dl)
  5. low high-density lipoprotein (HDL) cholesterol (<40 mg/dl in men and <50 mg/dl in women).
Sampling Method: Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Periprocedural myocardial injury (MI) | 24 hours after (percutaneous coroary intervention) PCI
  Periprocedural MI was defined as cardiac Troponin I release [5 times ULN] 24 hours after percutaneous coronary intervention

SECONDARY OUTCOMES:
Periprocedural myonecrosis | 24 hours after PCI
  Peri-procedural myonecrosis was defined as troponin I release of >1×ULN 24 hours after the intervention.

OTHER OUTCOMES:
inflammatory marker | 24 hours after PCI
  high sensitive C-reactive protein measurement 24 hours after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School Of Medicine, Department of Cardiology, Ankara, Turkey (Türkiye)